CLINICAL TRIAL: NCT03333603
Title: Pharmacokinetics and Safety Studies of Esomeprazole Use in Schizophrenic Patients
Brief Title: Pharmacokinetics and Safety Studies of Esomeprazole Use in Schizophrenia Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201601070MIND
Record Dates: First submitted 2017-01-17; First posted 2017-11-07 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2017-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Esomeprazole

STUDY DESIGN:
Intervention Model Description: Investigators will give 40 mg/day esomeprazole in the first two weeks and 80 mg/day from the third week to the end of the trial. Investigators will check the area under the concentration of metabolites of esomeprazoleon Day 1, Day 14 and Day 56 and the genotype of CYP2C19. The GI symptoms and related drug side effects will be evaluated.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- esomeprazole (Experimental): esomeprazole 40mg /tab oral Day1-Day14 then 40mg/2 tab oral Day15-Day56
  Interventions: Drug: esomeprazole

INTERVENTIONS:
Drug: esomeprazole — esomeprazole 40mg /tab oral Day1-Day14 then 40mg/2 tab oral Day15-Day56
  Other Names: Nexium

SUMMARY:
To evaluate the pharmacokinetic and safety for the esomeprazole use for schizophrenia

DETAILED DESCRIPTION:
Investigators prepare to recruit 30 schizophrenia patients in one year. Investigators will conduct a 8-week open label clinical trial for evaluation of the pharmacokinetic and safety of esomeprazole use for the schizophrenia. Investigators will give 40 mg/day esomeprazole in the first two weeks and 80 mg/day from the third week to the end of the trial. Investigators will check the area under the concentration of metabolites of esomeprazole on Day 1, Day 14 and Day 56 and the genotype of CYP2C19. The GI symptoms and related drug side effects will be evaluated.

ELIGIBILITY:
Inclusion criteria

1. 20-65 years old
2. Diagnosed as DSM-IV schizophrenia
3. No adjustment of dose of major antipsychotics for at least 4 weeks
4. Competence for inform consent

Exclusion criteria

1. Diagnosed with schizoaffective disorder or bipolar affective disorder or organic psychotic disorder
2. Meet the diagnostic criteria of any substance abuse or dependence in the past 6 months
3. History or evidence of any clinically significant medical or neurological disease, such as autoimmune disease, cancer, epilepsy, etc.
4. Mental retardation or pervasive developmental disorders
5. Past history of allergy to Esomeprazole
6. patient who is taking clozapine、 Depakin or Diazepam
7. Pregnant
8. The patient is under the order of involuntary admission

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration analysis | It will be assessed on Day 1 predose, Day 14 90 mins post dose, and Day 56 90 mins post dose
  The pharmacokinetic parameters for esomeprazole and its main metabolites

SECONDARY OUTCOMES:
CYP2C19 genotypes analysis | The genotype will be assessed on Day 1
  Investigators will genotype CYP2C19 genotype to determine that which metabolized type (poor metabolizer, intermediate metabolizer, and good metabolizer) of patients belong to.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Min Liu, Principal Investigator — Visiting Staff
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital Yunlin Branch, Taipei

IPD SHARING:
Plan to Share IPD: No